CLINICAL TRIAL: NCT02712814
Title: Subtypes of Provoked Vestibulodynia: A Prospective Study to Evaluate a Diagnostic Algorithm in Regard to Different Treatment Modalities
Brief Title: Subtypes of Provoked Vestibulodynia
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Ahinoam Lev-Sagie, MD, Meir Medical Center
Other Study IDs: 0152-15-COM1
Record Dates: First submitted 2016-03-05; First posted 2016-03-18 (Estimated); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Provoked Localized Vulvodynia
MeSH Terms: interventions — Estrogens; Low-Level Light Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Hormonally mediated PVD: * The entire vestibule is tender
  * The pain began while taking hormonal contraceptive
  * Secondary PVD
  * On exam, atrophic vestibular tissue (dry and thin)
  Interventions: Drug: Topical hormonal cream (estrogen)
- Congenital Neuroproliferative PVD: * The entire vestibule is tender
  * Primary PVD
  * There may be sensitivity to palpation of the umbilicus
  * Normal appearing vestibule
  Interventions: Procedure: Low Level Laser therapy
- Acquired neuroproliferative PVD: * The entire vestibule is tender
  * Secondary PVD, The pain had begun after a severe allergic reaction or vaginitis.
  * Normal appearing vestibule
  Interventions: Procedure: Low Level Laser therapy
- Hypertonic pelvic muscle dysfunction: * The pain is at 4-8 o'clock position of the vestibule with minimal or no pain in the upper vestibule
  * Pelvic floor muscles are tight and tender
  * Primary or Secondary PVD
  Interventions: Procedure: Pelvic floor physical therapy
- Neuroproliferative +Hypertonic: The entire vestibule is tender, but worse at 4-8 o'clock position of the vestibule
  * Primary PVD
  * There may be sensitivity to palpation of the umbilicus
  * Normal appearing vestibule
  * Pelvic floor muscles are tight and tender
  Interventions: Procedure: Pelvic floor physical therapy; Procedure: Low Level Laser therapy
- Hormonally +Hypertonic: The entire vestibule is tender, but worse at 4-8 o'clock position of the vestibule
  * The pain began while taking hormonal contraceptive
  * Secondary PVD
  * On exam, atrophic vestibular tissue (dry and thin)
  * Pelvic floor muscles are tight and tender
  Interventions: Drug: Topical hormonal cream (estrogen); Procedure: Pelvic floor physical therapy

INTERVENTIONS:
Drug: Topical hormonal cream (estrogen) — Patients will be instructed to stop hormonal contraception and to apply 0.1 ml topical cream containing 0.1% of estriol to the vestibule, once daily for 3 months
  Groups: Hormonally +Hypertonic; Hormonally mediated PVD
Procedure: Pelvic floor physical therapy — PF physical therapy once weekly for 3 months
  Groups: Hormonally +Hypertonic; Hypertonic pelvic muscle dysfunction; Neuroproliferative +Hypertonic
Procedure: Low Level Laser therapy — non-thermal laser irradiation (low levels of red and near infrared light) is applied directly to the vestibule
  Groups: Acquired neuroproliferative PVD; Congenital Neuroproliferative PVD; Neuroproliferative +Hypertonic

SUMMARY:
The proposed study will evaluate a clinical algorithm for the diagnosis and treatment of provoked vestibulodynia (PVD). The algorithm, distinguishes between four subtypes of PVD: hormonally mediated PVD, hypertonic pelvic floor dysfunction, congenital neuroproliferative PVD and acquired neuroproliferative PVD, based on a patient's history and physical exam. The study will follow patients diagnosed with PVD, for one year, and evaluate the treatment outcome in the different subgroups. Investigators hope that conducting a prospective study, showing clinical benefit and improved outcome for patients classified according to this method may change the common practice of "trial and error" based treatment, and will improve clinical results.

DETAILED DESCRIPTION:
Background Provoked vestibulodynia (PVD) is the term describing a syndrome of provoked, localized allodynia of the vestibule of the vulva, not explained by another condition, and lasting more than 3 months. PVD is not a defined disease but rather a symptom. It is thought that PVD represent a group of distinct disorders that have been classified together because they produce pain in the same anatomic location. Causes of these disorders include hormonal imbalance, mainly caused by hormonal contraception, nerve fiber proliferation in the vestibular mucosa and hypertonic pelvic floor dysfunction. PVD may appear with sexual debut or first attempts to insert a tampon (primary PVD) or can be a new onset of pain with activities that did not previously illicit pain (secondary PVD).

Studies found that different factors such as genetic, inflammatory mediators, recurrent vaginitis, allergy and trauma may be involved in the development of PVD. A high percentage of patients with vulvar pain report an antecedent history of vulvovaginal candida infection, although it is unknown if this represents a true increase in incidence or a misdiagnosis. It has been suggested that repeated vulvovaginal infections are a triggering event for some women leading to chronic vulvar pain. This observation has led to hypothesis that in patients with neurogenic vulnerability, an initiating event or series of events may lead to chronic vulvar pain.

Treatment of vulvodynia is generally predicated on a trial and error basis, because the pathogenesis is not defined. The result is that many forms of therapeutic interventions have been used, yet the evidence remains largely inconclusive, the response rate varies between 40-85%, and many women do not respond to any of the treatments. Unfavorable outcomes to therapy can be explained by grouping patients with different conditions under one diagnosis, and then studying an intervention that might only help one subset of the conditions. This can lead to an apparent lack of effect, due to dilution of the patient subpopulations.

A different approach to diagnosis and treatment of PVD was suggested by Dr. Andrew Goldstein. He classifies PVD into groups, based on history and examination findings:

1. Hormonally mediated PVD - The pain began while taking hormonal contraceptive or other medications that affect hormones, after removal of ovaries, breastfeeding or menopause. Typically, patients have a low calculated free testosterone and complain of dryness and decreased libido. The entire vestibule is tender and vestibular mucosa is often dry and thin. Treatment includes stopping hormonal contraception and application of topical estradiol with testosterone to the vestibule.
2. Hypertonic pelvic muscle dysfunction - In this subgroup, pelvic floor (PF) muscles become tight and tender. Patients often have other symptoms suggesting hypertonicity (urinary frequency, urgency and hesitancy, constipation, hemorrhoids and anal fissures), and predisposing factors, such as musculoskeletal disorders or anxiety may coexist. Typically, the pain is much worse at 4-8 o'clock position of the vestibule with minimal or no pain in the upper vestibule. Treatment includes PF physiotherapy, with an optional addition of muscle relaxants (valium suppositories and Botulinum toxin injections).
3. Neuroproliferative PVD- In this condition, women have an increased number of nociceptors in the vestibular mucosa. This group is further subdivided into congenital and acquired forms. In the congenital subgroup, vestibular pain has always been present, and there may be sensitivity to palpation of the belly button (which is an evidence of a congenital neuronal hyperplasia within the tissue derived from the urogenital sinus). With acquired neuroproliferative PVD, the pain may begin after a severe allergic reaction or vaginitis. There is tenderness of the entire vestibule. Treatments include topical anaesthetics, antidepressants, antiseizure drugs, capsaicin cream and vulvar vestibulectomy.

Goldstein's diagnostic algorithm is claimed to allow differentiation between different causes of PVD. In doing so, appropriate treatments to each subgroup can be selected, and their success rate should exceed the reported success rate in PVD treatment studies. Although investigators have a good personal experience with this method, the algorithm is not evidence based.

Objectives:

The proposed study is a prospective, cohort-based study, which will evaluate the characteristics of PVD-subgroups according to Goldstein's algorithm, patients' response to treatment and their outcome.

General aims: Define whether women that have been diagnosed according to Goldstein's algorithm experience higher rates of favorable outcome in comparison to those reported in the literature. This will allow us to study the effectiveness of this classification and to better define the subgroups.

Specific aims:

1. Describe the population of women with PVD attending the clinic, the distribution of criteria and the characteristics of women in each category.
2. Follow women diagnosed according to algorithm for one year and define treatment success.

Methods The proposed study is a prospective, cohort-based study. Patients will be recruited from the clinic for vulvovaginal disorders in Clalit Healthcare services in Jerusalem. The diagnostic procedures, patients' sub-classification and the proposed treatments in the current protocol are identical to those currently used in the clinic. Patients who fulfill diagnostic criteria of PVD and who will be willing to participate in the study will be asked to sign an informed consent and complete self-administered intake questionnaires requesting data about their PVD condition and its severity, various parameters of quality of life (QOL), general health, Ob\Gyn history, sexual function, psychometric characteristics (anxiety, depression etc) and demographics. After completing the questionnaires, each patient will undergo a standard evaluation, and will be diagnosed according to Goldstein's algorithm. Instructions for treatment will be given in regards to the diagnosis. Patients will be instructed to schedule follow-up appointments at 3,6,9, and 12 months. During follow-up appointments they will be assessed in regard to vestibular tenderness using various parameters, as well as by questionnaires of QOL and sexual function.

ELIGIBILITY:
Inclusion Criteria:

1. A history of 3 months or more of vulvar pain suggestive of PVD, i.e. symptoms of pain on vaginal penetration (insertional dyspareunia and/or pain with tampon insertion).
2. On exam, tenderness localized within the vestibule when being touched with a cotton-tip applicator.
3. No identifiable cause for the pain, such as vulvovaginal candidiasis, vaginal atrophy, desquamative inflammatory vaginitis (DIV), herpes, dermatitis or vulvar dystrophy.

Exclusion criteria:

1. other causes for vulvar pain
2. pregnancy or a planned pregnancy in the upcoming year
3. unprovoked or mixed vulvodynia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be recruited from the clinic for vulvovaginal disorders in Clalit Healthcare services in Jerusalem.
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Change of measure of Q tip test assesing pain intensity | Change in measure between recruitment to 3 months, 6 months 6 months, 9 months and 12 months
  The exam is performed by touching the vestibule with a cotton-tip applicator in 6 defined points (2,5,6,7, 10 and 12),while the patient is being asked to rate the intensity of pain verbally from 0 to 10 at each point.

SECONDARY OUTCOMES:
Visual analog scale (VAS) | Every 3 months for 1 year- 0, 3 months, 6 months, 9 months and 12 months
Measurement of vestibular tenderness using a vulvar algesiometer | Every 3 months for 1 year- 0, 3 months, 6 months, 9 months and 12 months
QOL parameters (questionnaire) | Every 3 months for 1 year- 0, 3 months, 6 months, 9 months and 12 months
Improvement in condition using a verbal report | Every 3 months for 1 year- 0, 3 months, 6 months, 9 months and 12 months
  in the follow-up appointments, patients will be asked to estimate the change in their condition, using percentage scaling: no or little improvement (<30%), moderate improvement (30-80%), much improvement (>80%) and total improvement (100%).
Tampon test | Every month for one year
  Patients will be provided with original Regular Tampax Tampons and will be instructed to deposit the tampon fully into the vagina above the level of the hymeneal ring with the applicator, remove the applicator from the vagina, and finally remove the tampon from the vagina by traction on the tampon string, immediately after vaginal insertion, without any lubrication. Patients will record the degree of pain during the entire insertion- removal experience, on a 0-10 pain numeric scale, with 0 meaning no pain, and 10 meaning the worst possible pain.
Female sexual function index | Every 3 months for 1 year- 0, 3 months, 6 months, 9 months and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ramat Eshkol Women health center, Clalit health Services, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No